CLINICAL TRIAL: NCT06040658
Title: Frailty Assessment in Vascular OUtpatients Review (FAVOUR Trial) - Comparing Feasibility and Prognostic Value of Commonly Used Assessments
Brief Title: Frailty Assessment in Vascular Hot Clinic Setting - Feasibility and Prognostic Value
Acronym: FAVOUR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Silje Welsh, Principle Investigator, University of Glasgow
Other Study IDs: GN23CE014
Record Dates: First submitted 2023-09-01; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Frailty; Frail Elderly Syndrome; Surgery
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vascular 'hot' clinic.: All adults (aged > 17 years) referred to an urgent-referral, consultant-led, Vascular Surgery outpatient clinic, who have capacity, will be eligible for inclusion in this study.
  Interventions: Diagnostic Test: Frailty assessment

INTERVENTIONS:
Diagnostic Test: Frailty assessment — Rockwood Clinical Frailty Scale
Diagnostic Test: Frailty assessment — Frail NonDisabled Questionnaire (FiND)
Diagnostic Test: Frailty assessment — Clinician's subjective 'end-of-bed' test
Diagnostic Test: Frailty assessment — Healthcare Improvement Scotland FRAIL Scale
Diagnostic Test: Frailty assessment — 11-item modified Frailty Index (mFI-11)

SUMMARY:
A single-centre prospective study of feasibility assessing the suitability of introducing routine frailty screening in a controlled, and reproducible, outpatient department setting for Vascular Surgery patients. This study will also perform head-to-head comparisons of the prognostic value of five frailty assessment tools, selected based on the previous demonstration of their popularity and familiarity within the speciality, their designs being based on different theories of frailty and that some are endorsed by local healthcare police. Inter-user variability (patient self assessment and clinician assessment will also be compared).

DETAILED DESCRIPTION:
This single-centre prospective cohort study of feasibility, is conducted in a rapid-referral vascular surgery clinic, serving a population of 2 million. Capax adults (>18years), attending clinic for any reason are eligible for inclusion. Five frailty assessments are completed at the clinic by patient (Rockwood Clinical Frailty Scale [CFS] and Frail NonDisabled Questionnaire [FiND]), clinician (CFS, Health care Improvement Scotland FRAIL Scale and 'Initial Clinical Evaluation') and researcher (11-item modified Frailty Index, mFI-11). Consistent with feasibility objectives, outcome measures include recruitment rates, frailty assessment completion rates, time-to-complete assessments and inter-rater variability. Electronic follow-up at 30-days and 1-year will assess home-time and mortality as prognostic indicators. Patients treated surgically/endovascularly will undergo additional 30-day and 1-year post-operative follow-up, outcome measures include: surgical procedure, mortality, complications (according to Clavien-Dindo Classification), length-of-stay, readmission rates, non-home discharge, home-time, higher social care requirements on discharge and amputation-free survival. Prognostic value will be compared by area under Receiver operator characteristic (ROC) curves. Continuous outcome variables will be analysed using Spearman's rank correlation coefficient. Inter-user agreement will be compared by percentage agreement in Cohen's Kappa coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 years or older)
* Attending Vascular Hot Clinic

Exclusion Criteria:

* Lacking capacity to provide informed consent
* Parent clinical team feel frailty assessment not suitable
* Non-English speaker without qualified translator present
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All referrals to vascular hot clinic are eligible for inclusion, preferentially recruiting new referrals. As frailty is related to age, but does not directly correlate with it, no age cut-off has been defined. As this is primarily a study of feasibility, patients will not be excluded/included based on presenting symptom or diagnosed pathology.
  A proxy (relative/friend/carer), if present, will also be invited to participate and assist with frailty assessments of the patients, where suitable. The participation of the proxy is dependent on the patient providing written consent agreeing to their participation, as well as the proxy being eligible to participate, according to the same inclusion/exclusion criteria set out for patients below.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing routine frailty assessment in a vascular clinic setting | During participant recruitment, over up to 4 months.
  Proportion of patients recruited (Number of recruited patients/[number of patients attending clinic - number of ineligible patients]).
Frailty assessment completion time | During participant recruitment, over up to 4 months.
  Time taken to complete assessments (presented in seconds). The less time taken, the better.
Frailty assessment completion rates | During participant recruitment, over up to 4 months.
  Proportion of assessments with non-completion. Calculated by: number of incomplete frailty assessments/total number of recruited patients, the lower the value the better.

SECONDARY OUTCOMES:
Assessing the prognostic value of selected frailty assessment tools (Home time - all patients) | 30-days and 1 year from recruitment/clinic attendance
  'Home time': this describes the number of full days at home (not as a hospital inpatient) over the follow up periods. All recruited patients will undergo this follow-up.
Assessing the prognostic value of selected frailty assessment tools (Mortality - all patients) | 30-days and 1 year from recruitment/clinic attendance
  Mortality: this will be calculated from date of recruitment. All recruited patients will undergo this follow-up.
Assessing the peri-operative prognostic value of selected frailty assessment tools (Mortality) | 30-days and 1 year from primary intervention offered following recruitment to study.
  For patients offered endovascular/surgical/hybrid intervention: mortality. Proportion of patients dead at follow up.
Assessing the peri-operative prognostic value of selected frailty assessment tools (Complications) | 30-days and 1 year from primary intervention offered following recruitment to study.
  For patients offered endovascular/surgical/hybrid intervention: post-operative complications (according to the Clavien-Dindo Classification).
Assessing the peri-operative prognostic value of selected frailty assessment tools (Length of stay) | 30-days and 1 year from primary intervention offered following recruitment to study.
  For patients offered endovascular/surgical/hybrid intervention: length of hospital stay (full days). Calculated as number of full days as inpatient following admission for index procedure.
Assessing the peri-operative prognostic value of selected frailty assessment tools (Readmission) | 30-days from primary intervention offered following recruitment to study.
  For patients offered endovascular/surgical/hybrid intervention: readmission rates (to any speciality). This will be calculated by the proportion of patients readmitted to hospital following index procedure/the number of patients undergoing surgical/endovascular treatment.
Assessing the peri-operative prognostic value of selected frailty assessment tools (Non-home discharge) | 30-days from primary intervention offered following recruitment to study.
  For patients offered endovascular/surgical/hybrid intervention: non-home discharge. This will be calculated by the proportion of patients who are discharged to place of residence differing from their preoperative residence/total number of patients undergoing surgical/endovascular treatment. For example, from private residence preoperatively to care home.
Assessing the peri-operative prognostic value of selected frailty assessment tools (Home time) | 30-days and 1 year from primary intervention offered following recruitment to study.
  For patients offered endovascular/surgical/hybrid intervention: home time. See outcome 4.
Assessing the peri-operative prognostic value of selected frailty assessment tools (Social care requirements) | 30-days from primary intervention offered following recruitment to study.
  For patients offered endovascular/surgical/hybrid intervention: discharge with a higher level of social care requirements. This will be presented as the proportion of patients discharged with greater social care requirements than before their index admission/'total number of patients offered surgical or endovascular treatment. E.g., a patient is admitted preopertively with three times daily package of care and discharged with four times daily package of care

CONTACTS AND LOCATIONS:
Overall Officials: Quinn, Study Director — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pseudonymised research data will be uploaded to appropriate data registry

REFERENCES:
- [Derived] Welsh SA, Hussey K, Brittenden J, Orr DJ, Quinn T. Frailty Assessment in Vascular OUtpatients Review (FAVOUR) protocol: single-centre prospective cohort study comparing feasibility and prognostic value of commonly used frailty assessment tools. BMJ Open. 2023 Dec 9;13(12):e079387. doi: 10.1136/bmjopen-2023-079387. PMID 38070914